CLINICAL TRIAL: NCT00508092
Title: Combined Nerve Blockade and Local Infiltration Anesthesia in Appendectomy - A Blinded Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Berkshire NHS Foundation Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q1602/168
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Pain, Postoperative
Keywords: appendicectomy; pain; local anaesthetic; nerve block; Post operative pain following appendicectomy
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): lanz incision appendectomy
  Interventions: Procedure: local anesthetic administration
- B (Active Comparator): lanz incision appendectomy
  Interventions: Procedure: local anesthetic administration

INTERVENTIONS:
Procedure: local anesthetic administration — Pre incision skin infiltration with local anesthetic 0.5% bupivacaine by weight
  OR
  Pre incision skin infiltration and deeper field infiltration (deep to external oblique) with local anesthetic 0.5% bupivavcaine by weight

SUMMARY:
The purpose of this study is to assess whether the use of local anesthetic to numb the nerves that run deeper in the abdominal wall gives better post operative pain control than just infiltrating local anesthetic to the wound edges.

DETAILED DESCRIPTION:
Local anesthetic is often administered during an operation to reduce post operative wound pain. Whilst this is frequently done during an appendectomy there is currently no evidence to suggest whether there is any benefit to the patient to injecting the local anesthetic deeper to block the nerves supplying abdominal wall sensation, compared to using it just in the skin around the wound.

Comparison: Post operative pain scores following appendectomy for patients given skin infiltration of local anesthetic (pre incision), compared to patients given both preincision wound infiltration and deeper field infiltration with local anesthetic(deep to external oblique).

ELIGIBILITY:
Inclusion Criteria:

* Lanz incision appendectomy as starting procedure, including those where an alternative cause for symptoms is found at operation and those where incision is later extended/changed (these may be sub grouped at time of analysis)
* Consent obtained

Exclusion Criteria:

* Laparoscopic appendectomy
* Appendectomy at time of laparotomy/other incision

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Post operative pain score | 1 hour, 4 hours, 8 hours, 24 hours and on discharge

SECONDARY OUTCOMES:
Post operative nausea and vomiting | 1 hour, 4 hours, 8 hours, 24 hours and on discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan K Randall, MRCS, Principal Investigator — Royal Berkshire NHS Foundation Trust; Simon B Middleton, FRCS, Study Chair — Royal Berkshire NHS Foundation Trust; Arnold Goede, MRCS, Study Director — Royal Berkshire NHS Foundation Trust
Locations (1):
- Royal Berkshire Hospital, Reading, Berkshire, United Kingdom